CLINICAL TRIAL: NCT05768984
Title: The Effect of an Empowerment Program on Ruminative Thoughts, Fatigue, and Psychological Resilience of Cancer Survivors
Brief Title: Empowerment Program for Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinem Ocalan (Other)
Responsible Party: Sponsor-Investigator, Sinem Ocalan, Research assistant, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA-22037
Record Dates: First submitted 2023-02-28; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cancer Survivors
Keywords: Patient; Nursing; Cancer; Psychological resilience; Rumination; Fatigue
MeSH Terms: conditions — Neoplasms; Rumination Syndrome; Fatigue

STUDY DESIGN:
Intervention Model Description: Permission will be taken from Hacettepe University Oncology Hospital for the research. However, due to the pandemic conditions, to protect the health of both researchers and participants, group studies were moved to the online platform and the sessions were planned as online (zoom sessions). The sample size of the study was calculated with the G-Power 3.1 program. Since a similar study could not be found in the literature, it was determined that the sample should consist of 56 people, 28 in the intervention group and 28 in the control group, by calculating with .80 power and .05 error level, based on the medium effect size for the .25 variance analysis suggested by Cohen. However, it is foreseen that it would be appropriate to reach 10% more people (Total 62) of the total number calculated considering that there may be a loss of participants during the process and to be participants in the 31 intervention and 31 control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Empowerment program will be implemented.
  Interventions: Other: Empowerment program
- Control group (No Intervention): No program will be implemented.

INTERVENTIONS:
Other: Empowerment program — It is planned to conduct the empowerment program online (zoom session). For this, to protect each individual's privacy, a quiet, bright and ventilated, spacious physical environment and technological elements such as computers, headphones, microphones and internet connection are needed. The empowerment program was planned as a total of 10 sessions, one session per week. In the program, goals and objectives have been established for each session. These aims and objectives will be shared with the participants before each session. The application time of each session is planned as an average of 90 minutes.
  Arms: Experimental group

SUMMARY:
This study aims to decrease cancer survivors' intrusive ruminative thoughts and cancer-related fatigue and increase their purposive ruminative thoughts and psychological resilience. In this context, an online (Zoom) 10-session empowerment program based on the literature will be implemented for cancer survivors.

DETAILED DESCRIPTION:
From the time they were diagnosed with cancer, individuals struggle with ruminative thoughts about why they have this disease, whether they will get better during the treatment process, whether the disease will recur in the future, and cognitive, physical, and emotional fatigue, the cause of which cannot be fully explained. All these processes continue to negatively affect the lives of cancer survivors during the remission period. Studies show that when cancer survivors manage this stressful process well and learn effective coping methods, they can come out of it by developing their psychological resilience. Therefore, this study aimed to determine the effect of an empowerment program to be applied to cancer survivors' ruminative thoughts, cancer-related fatigue, and psychological resilience.

The hypotheses of this research are:

H 1-1: There is a difference between ruminative thinking scores at the end of the empowerment program applied to individuals with cancer in remission and in the follow-up measurement compared to the pre-program and control groups.

H 1-2: There is a difference between cancer-related fatigue scores at the end of the empowerment program applied to individuals with cancer in remission and in the follow-up measurement compared to the pre-program and control groups.

H 1-3: There is a difference between psychological resilience scores at the end of the empowerment program applied to individuals with cancer in remission and in the follow-up measurement compared to the pre-program and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being between the ages of 18-65,
* To have knowledge of reading and writing in Turkish,
* Being in remission
* To have technical equipment (camera, microphone, computer) and usage knowledge to participate in the online group session

Exclusion Criteria:

- To have received psychological support in the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Event-Related Rumination Inventory at day 70, and day 160 | day 0, day 70, and day 160
  It was developed by Cann et al. (2011). The 20-item scale has subscales to evaluate two forms of rumination, "intrusive" and "deliberate". The first ten items measure intrusive rumination, and the second ten items measure deliberate rumination. Each item in the scale is in a 4-point Likert type and is scored as 0 = never, 3 = often. There is no total score in this scale, but subscale scores reveal rumination scores. Scores on each subscale range from 0 to 30. High scores obtained from each sub-dimension of the scale indicate the existence of a ruminative thought tendency towards the said dimension.
Change from Baseline Cancer Fatigue Scale at day 70, and day 160 | day 0, day 70, and day 160
  It was developed by Okayama et al. in 2003. Consisting of 15 items, the scale has a 5-point Likert type ranging from 'no' (1) to 'too much' (5). It consists of three sub-dimensions: physical (items 1,2,3,6,9,12,15), emotional (items 5,8,11,14), cognitive (items 4,7,10,13). . The range of scores to be taken from the scale is between 0 and 28 points for the physical subscale, and 0 to 16 points for the emotional and cognitive subscale. Total fatigue is the sum of these subscale scores and the maximum total score is 60. The higher the total score, the more severe the fatigue is considered.
Change from Baseline Connor-Davidson Resilience Scale at day 70, and day 160 | day 0, day 70, and day 160
  It was developed by Connor and Davidson (2003). The 25-item scale is in a 5-point Likert structure as 'not at all true' (0) and 'always true' (4). The scale consists of 3 subscales: 'Perseverance and Personal Efficiency' (15 items), 'Resistance to Negativity' (6 items) and 'Tension to Spirituality' (3 items). The lowest and highest values vary between 0-100, and the higher score obtained from the scale indicates greater psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Öcalan, Res. Asist., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No